CLINICAL TRIAL: NCT05121090
Title: Prevention of Child Obesity: an Interventional Study of a Personalized Multidisciplinary Care Efficacy in Children of Primary School
Brief Title: Lille Study for Childhood Health Promotion
Acronym: ELIPSE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: National Center for Precision Diabetic Medicine,PreciDIAB (Unknown); PrevSanté MEL (Unknown); APESAL (Unknown); National Research Agency, France (Other); European Union (Other); Hauts-de-France Regional Council (Unknown); University of Lille Nord de France (Other); Groupement des Hôpitaux de l'Institut Catholique de Lille (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020_43; 2020-A02217-32 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-09-23; First posted 2021-11-16 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Overweight, Infant; Overweight and Obesity; Overweight, Childhood
Keywords: Paediatric overweight and obesity; Childhood obesity; Personalized prevention and medicine; Educational program; Genetic of obesity
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Educational program — The educational program is based on dietary, physical activity, psychology, and sophrology approaches dispensed by health care professionals. Evaluations will consist of anthropometric measurements (height, weight, body mass index), behavioural questionnaires, and basic physical tests (handgrip, squats, balance, …).
  Optionally, a saliva collection will be proposed to obtain the DNA required for genetic analyses.

SUMMARY:
Obesity could be avoided but once declared it become a chronic disease with numerous health complications, including cardiovascular and metabolic diseases, cancers, and finally a loss of life expectancy. Considering that after the age of 6 years old, half of the obese children will become obese adults, the WHO has been declared childhood obesity prevention as a health priority area. Large-scale prevention of obesity is challenging and it would be more efficient to proceed to early identification of high risks children to implement personalized prevention.

The ELIPSE study main objective is to evaluate the efficacy of personalized multidisciplinary care to reduce the BMI of overweight or obese children. A 2 years educational program will be evaluated at short and longer terms (after a 12 months follow-up), and its benefits will also be assessed based on comparison with a historical control group.

Along with efficacy evaluation, scientific objectives were designed to investigate clinical, genetic, social, and behavioural risk factors and to analyse potential correlations between these factors and a predisposition to overweight or obesity. Moreover, advanced analyses will be performed to decipher the impact of diverse risk profiles on the efficacy of the educational program.

The motive of the ELIPSE study is to promote the health and well-being of children and their families to tackle the health burden represented by childhood overweight and obesity. Combined with innovative scientific objectives, this study ambitions to develop more efficient and more personalized preventive care methods.

ELIGIBILITY:
Inclusion Criteria:

* Children from the first year of primary school in Lille City
* Overweight or obese children as defined by the IOTF and/or with at least one of the following risk factors: 1) early adiposity rebound (before 6 years old), 2) an upward crossing of major percentiles on the BMI curve (after 6 years old).
* Children whose legal tutor(s) is(are) able to understand the enlightened information.
* Children whose legal tutor(s) has(ve) signed the free and informed consent.

Exclusion Criteria:

* Refusal from children or their tutors to participate in the study.
* Impossibility to participate in the study in its totality.
* Pathology known to impact the BMI: follow-up care for eating behaviour problems, endocrine disorders (hypercorticism, hypothyroidism, growth factor deficiency, hypothalamic-hypophysis lesions), genetic disorders (Prader Willi syndrome, Bardet-Biedl syndrome), drugs that affect body weight (antidepressant, neuroleptics, corticoids).
* Previous participation in a similar educational program.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from the first year of primary school in Lille City
Sampling Method: Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in BMI Z-score | At the end of the educational program, an average of 2 years after inclusion
  The objective is to estimate the mean variation of the BMI Z-score between the inclusion and the end of the educational program, after 2 years.
  Body mass index z score is based on previous results, estimate that the BMI Z-score will be decreased by 0.3 +/- 0.6 SD.

SECONDARY OUTCOMES:
BMI Z-score between children included in the study and a historical control group | At the end of the educational program, an average of 2 years after inclusion
  At the end of the educational program (2 years after inclusion), BMI Z-scores of children who completed the study will be compared to those of a historical control group composed of children of similar ages who did not benefit from an educational program
Changes in BMI Z-score. | At the end of the educational program follow-up, an average of 3 years after inclusion
  The objective is to estimate the mean variation of the BMI Z-score between the inclusion and the end of the educational program follow-up, 3 years after inclusion.
Correlation between clinical and environmental variables and changes in BMI Z-score | At the end of the educational program, an average of 2 years after inclusion
  The objective is to study the statistical relationship between the BMI Z-score and clinical and environmental variables: birth weight (kg), mother's BMI (kg/m^2), gestationnel diabetes, parental weight loss surgery, number of child(ren) in the family, socioeconomic status evaluated by the parents socio-professional category (french indices), smoking during pregrancy)
Impact of polygenic risk scores of obesity on changes in BMI Z-score | Through study completion, an average of 3 years after inclusion
  A multi-variants analysis will be performed using DNA chips to identify loci associated with an increase of the BMI to obtained a polygenic risk score. This score will then be included as a variable for the analyses of the secondary outcome
Impact of rare pathogenic mutations causing obesity on changes in BMI Z-score. | Through study completion, an average of 3 years after inclusion
  A whole-exome sequencing will be performed, followed by the identification of rare mutations involved in obesity or novel genes

CONTACTS AND LOCATIONS:
Overall Officials: Louise Montagne, MD, Principal Investigator — Lille Catholic University